CLINICAL TRIAL: NCT05333484
Title: Effects of a 12-week Pilates Program on Basal Metabolic Rate, Body Composition, Physical Activity in Middle-aged and Elder Females
Brief Title: 12-week Pilates Program on Community-dwelling Middle-aged Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Wen Ching Huang, Associated Professor, National Taipei University of Nursing and Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMHIRB-102001
Record Dates: First submitted 2022-03-29; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Functional Fitness; Health Promotion; Exercise; Frail Elderly Syndrome
Keywords: Pilates; middle-aged women
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The study was quasi-experimental design with a parallel control group and the participants were recruited with convenience sampling method.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates Intervention Group (Experimental): 12-week programed Pilates intervention
  Interventions: Other: Programed Pilates
- Control Group (No Intervention): maintenance of normal lifestyle in control group

INTERVENTIONS:
Other: Programed Pilates — The 60 min Pilates sessions were held twice a week for 12 weeks. Each session included three stages: 10 min of warm-up exercises, 40 min of floor-based Pilates training, and 10 min of cool-down exercises. Each stage was adjusted according to the participants' physical capacity. Only participants with an attendance rate of > 80% were included in the final sample. The content of the exercise program was determined according to their muscular strength, flexibility, and fitness levels. The training course was divided into three levels: elementary, intermediate, and advanced. Each motion was performed in conjunction with a specific breathing pattern for effective muscle activations of each exercise.
  Arms: Pilates Intervention Group

SUMMARY:
The purpose of this study was to investigate the effects of a Pilates exercise intervention program on functional physical fitness in community-dwelling middle-aged women.

DETAILED DESCRIPTION:
Based on quasi-experimental design with a parallel control group, Subjects were allocated into to intervention group and control group with convenience sampling method. The primary outcome included body composition, basal metabolic rate, and functional physical fitness-comprising cardiovascular capacity (3-minute step test), flexibility (sit-and-reach test), muscular strength of upper limbs (grip-strength test), muscular strength of lower limbs (30 s chair stand test), core strength (bent-knee sit-up test), agility (8-foot timed up-and-go test), static balance (single-leg stance with eyes closed test), and dynamic balance (functional reach test), assessed in both groups before and after the 12-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* Female 45-64 years old in age

Exclusion Criteria:

* cognitive-function impairment
* spinal disease
* unsuitability for engaging in physical activity (e.g., because of severe cardiovascular disease)
* muscular strength affected by medication for nervous system diseases.

Ages: 45 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
The effects of 12-week Pilates program on body-fat and muscular percentage measured by Physion-XP | 12 weeks
  The body composition is simultaneously measured by Physion-XP for outcome measures including body-fat percentage (%), and muscular percentage (%) in the upper and lower limbs. The higher muscular percentage and lower body-fat percentage would be associated with appropriate fitness. Changes of body-fat percentage, and muscular percentage in the upper and lower limbs measures will be assessed at the 0 week, and 12 weeks.
The effects of 12-week Pilates program on weight measured by height scale | 12 weeks
  The body weight (kilograms) is measured by height scale. The higher body weight would be associated with obesity and the he lower weight without diseases and medical conditoins means the better fitness. Changes of body weight measures will be assessed at the 0 week, and 12 weeks.
The effects of 12-week Pilates program on height measured by height scale | 12 weeks
  The height (meters) is measured by height scale. The higher height would be associated with body growth. Changes of height measures will be assessed at the 0 week, and 12 weeks.
The effects of 12-week Pilates program on BMI calculated by height and weight | 12 weeks
  The Body Mass Index (BMI) is calculated by weight and height measures. Body Mass Index is a simple calculation using a person's height and weight. The formula is BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in meters squared. The higher BMI would be associated with obesity. Changes of BMI measures will be assessed at the 0 week, and 12 weeks.
The effects of 12-week Pilates program on basal metabolic rate measured by MedGem Indirect Calorimeter | 12 weeks
  The handheld MedGem Indirect Calorimeter is used to measure basal metabolic rate. The higher outcomes mean the higher basal metabolic rate. Changes of basal metabolic rate will be assessed at the 0 week, and 12 weeks.
The effects of 12-week Pilates program on cardiovascular capacity | 12 weeks
  The cardiovascular capacity is evaluated by 3-minute step test. The higher index of cardiovascular capacity means the higher cardiovascular fitness. Changes of cardiovascular capacity will be assessed at the 0 week, and 12 weeks.
The effects of 12-week Pilates program on flexibility | 12 weeks
  The flexibility is evaluated by sit-and-reach test. The longer distance of test means the higher flexibility fitness. Changes of flexibility will be assessed at the 0 week, and 12 weeks.
The effects of 12-week Pilates program on muscular strength of upper limbs | 12 weeks
  The muscular strength of upper limbs is evaluated by grip-strength test. The higher strength of test means the higher strength fitness in upper limbs. Changes of muscular strength of upper limbs will be assessed at the 0 week, and 12 weeks.
The effects of 12-week Pilates program on muscular strength of lower limbs | 12 weeks
  The muscular strength of lower limbs is evaluated by 30 s chair stand test. The higher repetitions mean the higher strength fitness in lower limbs. Changes of functional physical fitness will be assessed at the 0 week, and 12 weeks.
The effects of 12-week Pilates program on core strength endurance | 12 weeks
  The core strength endurance is evaluated by 1-minute bent-knee sit-up test. The higher repetitions mean the higher core strength endurance fitness. Changes of core strength endurance will be assessed at the 0 week, and 12 weeks.
The effects of 12-week Pilates program on agility | 12 weeks
  The agility is evaluated by 8-foot timed up-and-go test. The shorter time for the task means the higher agility fitness. Changes of agility will be assessed at the 0 week, and 12 weeks.
The effects of 12-week Pilates program on static balance | 12 weeks
  The static balance is evaluated by single-leg stance with eyes closed test. The longer time for single-leg stance with eyes closed means the higher static balance fitness. Changes of static balance will be assessed at the 0 week, and 12 weeks.
The effects of 12-week Pilates program on dynamic balance | 12 weeks
  The dynamic balance is evaluated by functional reach test. The longer distance reach with stability means the higher dynamic balance fitness. Changes of dynamic balance will be assessed at the 0 week, and 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Ching Huang, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Camillians Saint Mary's Hospital Luodong, Yilan, Taiwan